CLINICAL TRIAL: NCT02259556
Title: CD30-directed Chimeric Antigen Receptor T (CART30) Therapy in Relapsed and Refractory CD30 Positive Lymphomas
Acronym: CART30
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-011
Record Dates: First submitted 2014-10-05; First posted 2014-10-08 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-CD30 CAR T cells (Experimental): Patients receive CART30 cell infusions with an escalation dose.
  Interventions: Biological: CART30

INTERVENTIONS:
Biological: CART30 — Cells will be infused 1 day after the completion of conditioning regimen.
  Other Names: anti-CD30 CAR T cells

SUMMARY:
Chimeric antigen receptor-modified T cells (CART) holds great promise for treatment of tumors. In this trial, CD30 positive Hodgkin's lymphoma and Non-Hodgkin's lymphoma will be treated by CD30-specific CART cells (CART30).

DETAILED DESCRIPTION:
When patients enroll on this trial, autologous CART-33 cells were generated from the mononuclear cells of 50 to 90 ml of the patient's peripheral blood (PB). During the term of cell preparation of CART30, patients will receive a conditioning regimen including cyclophosphamide and fludarabine. One day after completing conditioning regimen, the patient will be given infusions of CART30 cells into the vein in escalating doses over a period of 3 to 5 consecutive days.

Extra blood will be drawn to measure the persistence of CART30 in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with CD30+ Hodgkin lymphoma and Non-Hodgkin lymphoma relapsing after autologous stem-cell transplantation (ASCT), or refractory to 2 multidrug regimens and/or anti-CD30 antibody treatment.
* Newly diagnosed CD30+ Hodgkin lymphoma and Non-Hodgkin lymphoma patients who are unable to receive or complete standard chemotherapy.
* Karnofsky or Lansky score greater than 60%.
* Expected survival>12 weeks.
* Creatinine<2.5mg/dl.
* ALT (alanine aminotransferase)/AST (aspartate aminotransferase)<3 fold normal.
* Bilirubin<2.5mg/dl.
* Pulse oximetry of >90% on room air.
* Adequate pulmonary function with FEV1, FVC and DLCO greater than or equal to 50% of expected corrected for hemoglobin.
* Available autologous T cells with 10% or more expression of CD30 CAR determined by flow-cytometry.
* Patients or legal guardians must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects. Patients or their guardians will be given a copy of the consent form.

Exclusion Criteria:

* Active infection such as hepatitis B or C.
* Receive anti-CD30 antibody-based therapy within recent 6 weeks.
* Current use of systemic corticosteroids.
* Pregnant or lactating.
* Confirmed tumor in pulmonary and archenteric tissues.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of related adverse events | untill week 24

SECONDARY OUTCOMES:
Anti-tumor response to CART30 cell infusions | Up to 24 weeks
  Evaluated mainly by computed tomography scanning

OTHER OUTCOMES:
in vivo existence of CART30 | 1 year
  Measure mainly by the changes of CAR molecule levels in blood

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Ph.D, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China